| NCT number: NCT03279692 |
|-------------------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates



OHRS 02.03.2017

**Protocol Title:** Phase II Trial of Pembrolizumab in Recurrent or Residual High Grade Meningioma

#### DF/HCC Principal Research Doctor / Institution:

Priscilla Brastianos, MD / Massachusetts General Hospital

#### DF/HCC Site-Responsible Research Doctor / Institution:

Eudocia Karem Quant Lee, MD, MPH / Dana-Farber Cancer Institute

Main ICF

#### A. INTRODUCTION

You are invited to take part in a clinical trial, a type of research study, because you have Recurrent or Residual High Grade Meningioma. This research study is studying a drug as a possible treatment for this diagnosis.

The name of the study drug involved in this study is Pembrolizumab

For purposes of this research, you will be referred to as a "participant".

It is expected that about 26 people will take part in this research study.

Merck, a pharmaceutical company, is supporting this research study by providing funding for the research study, including the study drug.

Dana-Farber Cancer Institute has a financial interest in the investigational compound used in this trial, Pembrolizumab, which may be affected by the outcome of this research. The Institute has taken steps to manage any conflict of interest created by this financial interest. Additional information is available in the Patient Information Sheet available to participants.

This research consent form explains why this research study is being done, what is involved in participating in the research study, the possible risks and benefits of participation, alternatives to participation, and your rights as a research participant. The decision to participate is yours. If you decide to participate, please sign and date at the end of this form. We will give you a copy so that you can refer to it while you are involved in this research study. If you choose not to


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | A-85 |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

participate in this research study, the research doctors will discuss other treatment options with you and/or refer you back to your primary doctor. We encourage you to take some time to think this over, to discuss it with other people and your primary doctor, and to ask questions now and at any time in the future.

## B. WHY IS THIS RESEARCH STUDY BEING DONE?

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for your specific disease but it has been approved for other uses.

In this research study, we are studying pembrolizumab in participants with meningioma. Research studies have shown that meningioma tumor cells express a gene called PD-L1. We will be looking to determine whether the study drug may stop this gene from being activated on your tumor and whether the study drug may stop the tumor cells from growing.

## C. WHAT OTHER OPTIONS ARE THERE?

Taking part in this research study is voluntary. Instead of being in this research study, you have other options which may include the following:

- Receive standard treatment including radiation or surgery
- Take part in another research study.
- Receive no therapy specific to your cancer.
- Comfort care, also called palliative care. This type of care may help to reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to treat the symptoms.

Please talk to the research doctor about your options before you decide whether you will take part in this research study.

#### 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | VVC) 5-88 (Mc), WI |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

#### D. WHAT IS INVOLVED IN THE RESEARCH STUDY?

Sometimes it is hard to keep track of all of the details and procedures that are part of a research study. We will describe them in this consent form and you can refer to this at any time during the research study.

#### Before the research starts (screening):

After signing this consent form, you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

- A medical history, which includes demographics, questions about your health, current medications, and any allergies.
- Physical exam, including measurements of your vital signs and weight.
- Performance status, which evaluates how you are able to carry on with your usual activities.
- An assessment of your tumor by MRI (Magnetic Resonance Imaging)
  unless you have extracranial metastases (cancer that has spread from
  your tumor to a different part of your body) in which a CT (Computerized
  Tomography) scan of your chest, abdomen, and pelvis will be performed
  as well.
- **Blood tests**, approximately 2 tablespoons of blood will be collected at the study visits for research and clinical purposes.
- Your previously collected and stored tissue (archival tissue) will be obtained for tests. No additional tissue will be collected.

If these tests show that you are eligible to participate in the research study, you may begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

#### **Study Treatment Overview:**


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | - 55 Aug 10 A |

| 3/2 | 180 | 20 | 23 | 4:3 | 5 | PM |
|------|-----|----|----|------|---|-------|
| VI 4 | | 20 | | T. U | J | - IVI |

| NCT | number: NCT03279692 |
|-----|---------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

 Infused Study Drug: You will be given pembrolizumab once every cycle.
 Each cycle lasts 21 days. You will be given this study drug into your vein (by intravenous infusion) over about 30 minutes.

#### Research Study Plan:

| | | | D | | Treatm | ent Cycle | S | | | End of | 9 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | 4 | 2 | 2 | 1 | To be re | epeated | beyond | 8 cycles | End of | Follow-Up |
| | | | 2 | 3 | 4 | 5 | 6 | 7 | 8 | Treatment | |
| Medical History | X | | | | | | | | | | |
| Physical Exam | | X | X | X | X | X | X | X | X | X | X |
| Performance Status | | X | X | X | X | X | X | X | X | X | X |
| Tumor Assessment | X | | | X | | X | | X | | X | |
| Blood Tests | Х | X | X | X | X | X | X | X | X | X | |
| Archival Tissue | X | | | | | | | | | | |
| Pembrolizumab | | X | X | X | X | X | X | X | X | | |

#### Planned Follow-up:

If you decide to stop the study drug and your disease has not gotten worse we would like you to come into the clinic once every 6 weeks for a MRI or CT scan until you either start a new anti-cancer treatment, your disease gets worse, or the end of the study, whichever comes first.

If you are taken off of the study we would like to follow up with you every 3 months either through scheduling a clinic visit or reviewing your medical record. Keeping in touch with you and checking your condition helps us look at the long-term effects of the research study.

# E. How long will I be in this research study?

You will be in this research study for as long as you are responding to and tolerating treatment.

You may be taken off the research study drug for many reasons including if:

- It is considered to be in your best interest
- The study treatment or procedures are found to be unsafe or ineffective
- There is any problem with following study treatments and procedures
- You are a female and become pregnant or plan to become pregnant 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

- Your condition worsens
- A decision is made to close the study
- Or for other unforeseen reasons that make it necessary to stop your participation in the research study

If you are removed from the research study, the research doctor will explain to you why you were removed.

In addition, you can stop participating in the research study at any time, however, the FDA requires that any information collected up to the point of your withdrawal cannot be removed from the study. If you decide to stop participating in this research study, we encourage you to talk to the research doctor and your primary doctor first.

#### F. WHAT ARE THE RISKS OR DISCOMFORTS OF THE RESEARCH STUDY?

There are risks to taking part in any research study. One risk is that you may get a study drug that does not help treat your disease or that makes your condition or disease worse. Another risk is that there may be side effects.

All cancer treatments can have side effects, which can range from mild and reversible to severe, long lasting and possibly life-threatening. There is a great deal of variability among side effects of different cancer treatments and between individuals. In a research study, all of the risks or side effects may not be known before you start the study. You need to tell your doctor or a member of the study team immediately if you experience any side effects.

Everyone in the research study will be watched carefully for side effects. You will be monitored during the administration of study drugs to keep track of your blood counts and organ function, particularly your kidney and liver function. If you experience side effects, they may go away after you stop taking the study drug. Some side effects can be mild; but others can be long lasting and may never go away. Some may be life-threatening or fatal.

Since the effect of the study drug(s) taken with other medications may not be known, it is important that you tell the research doctor about all prescription and non-prescription drugs, herbal preparations and nutritional supplements that you are taking or planning to take. There may also be some foods that you should


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | 5000 0.88 0501. 99 |

| 3 | 128 | 120 | 123 | 4:35 | PM |
|---|-----|-----|-----|------|---------|
| • | 720 | 124 | | T.UU | , I IVI |

| NCT number: NCT03279692 |
|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

avoid while on this research study and your research doctor will review this information with you.

During the research study, you will be notified of newly discovered side effects or significant findings, which may affect your health or willingness to participate. You may be asked to sign a new consent form that shows that you have been informed of new information relating to this research study.

#### Risks Associated with pembrolizumab:

### Very common (at least 20% chance that this will happen):

- · Itching of the skin
- Diarrhea (this may be associated with a more serious inflammatory condition)
- Cough (this may be associated with a more serious inflammatory condition)
- Rash
- Fatigue

#### Common (Between a 10-20% chance that this will happen):

- Joint pain
- Fever. This may be serious or life threatening.
- Back pain

#### Occasional (between a 1% to a 10% chance that this will happen):

- Too little thyroid hormone that controls how the body uses energy
  which may cause you to feel tired, gain weight, feel cold, and have
  infrequent or hard bowel movements. This may manifest as a serious
  immune-mediated side effect in 1% or fewer patients. (hypothyroidism)
- Too much thyroid hormone that controls how the body uses energy
  which may cause you to feel anxious, angry, weak, and tired, and may
  cause trembling, weight loss, hair loss, increased sweating, diarrhea,
  and difficulty sleeping. This may manifest as a serious immunemediated side effect in 1% or fewer patients. (hyperthyroidism)
- Inflammation of the lungs which may cause shortness of breath and cough. This may manifest as serious in 1% to 4% of patients and there is a rare chance that this may become life threatening. (pneumonitis)
- Inflammation of the large intestine (bowels/gut) which may cause stomach pain with loose or watery stools. This might manifest as serious in 1% to 4% of patients. (colitis)


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | |

| 3/2 | 8/202 | 3 4:35 | PM |
|-----|-------|--------|----|
|-----|-------|--------|----|

| NCT number: NCT03279692 |
|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

- Inflammation of the skin so you may have peeling of the skin, itching, and skin redness. In 1% or fewer patients this may cause widespread peeling of the skin. Rarely, this might become severe and life threatening, and involve the inside of the mouth, surface of the eye and genital area and/or may cause the top layer of your skin to peel from all over your body which can cause severe infection. (Stevens Johnsons Syndrome)
- Stomach cramps, pain in the abdomen due to cramping
- Loss of skin color and hair color (vitiligo)
- Low levels of salt in the blood, which can cause confusion, headaches, fatigue, muscle cramps, and make you feel sick to your stomach.
- Dizziness or fainting (low blood pressure), flushing, rash, fever, shortness of breath or sick to your stomach at the time of receiving your infusion (IV) or just after, or pain at the site of infusion. This may manifest as serious in less than 1% of patients and there is a rare chance that this may become life threatening.
- Arthritis, which is swelling of the joints.

# Rare but serious immune-mediated side effects (1% or less chance that this will happen):

- Inflammation of the liver which may cause you to feel not hungry, tired, have a mild fever, muscle or joint aches, nausea and vomiting, stomach pain, yellow eyes and skin, and dark urine. This may become serious or life threatening (hepatitis)
- Inflammation of the pituitary gland which may cause headaches, stomach discomfort, change in eyesight (double vision), change in behavior, few to no menstrual cycles (for women), weakness, vomiting, and dizziness or fainting (hypophysitis)
- Inflammation of the glands on top of the kidneys (adrenal glands)
  leading to insufficient hormone production causing tiredness, weight
  loss, muscle weakness, feeling faint, joint, muscle and abdominal
  aches, nausea, vomiting, loose or watery stools, fever, salt craving, and
  sometimes darkening of the skin like a suntan
- Inflammation of the kidney which may cause you to pass less urine, have cloudy urine, have blood in your urine, have swelling and lower back pain
- Inflammation of the muscles which may cause weakness or pain in the muscles

#### 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | A-85 |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

- Inflammation of the pancreas causing pain in the upper abdomen. This
  could cause nausea and vomiting that gets worse when you eat.
  (pancreatitis)
- Inflammation of the eye causing redness of the eye, blurred vision, sensitive to light, eye pain, see floaters or have headaches (uveitis)
- A condition when you may have too much sugar in your blood, may feel thirsty, and are likely to need regular insulin shots for treatment (diabetes).
- Inflammation of the nerves that may cause pain, weakness or tingling in the hands and feet, and may spread to the legs, arms, upper body leading to severe muscle weakness and possible temporary paralysis. This may become serious or life threatening.
- Inflammation of the heart muscle (myocarditis) that may cause your heart to have difficulty pumping blood throughout your body. This may cause chest pain, shortness of breath, and swelling of the legs. You may experience a fast or irregular heart rate causing dizziness or fainting. This might become severe, require hospitalization, and sometimes this condition can lead to death.
- A condition where you will feel weakness and fatigue of your hip and thigh muscles and an aching back caused by your body's immune system attacking your healthy cells and tissues. (polymyositis)
- Inflammation of the stomach and/or intestines which may result in bleeding, diarrhea, and perforations. This may be serious or life threatening. (gastroenteritis)

Some drug reactions can rarely be fatal and may occur even after discontinuation of pembrolizumab therapy.

Cancer research often includes biopsies, scans, x-rays that are also provided as routine care. The following describes the side effects of procedures done only for the purposes of research.

#### Risks Associated with MRI Scans:

When having an MRI (Magnetic Resonance Imaging) scan, you will lie still on a table that slides into a tunnel slightly wider than your body. People who feel uncomfortable in confined spaces (claustrophobia) may feel uncomfortable in the narrow cylinder. If you feel uncomfortable in confined spaces, please tell your research doctor. Your doctor may give you a medication to make you feel more comfortable. As images are taken, a loud banging noise will be produced.


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

Earplugs or headphones will be available if needed. The MRI can be stopped at any time at your request, but the scan may not be complete.

#### Risks Associated with Contrast Agents Used During Scans:

There is a small risk with using a contrast agent that is injected into a vein during the MRI. The contrast agent is a special dye that highlights organs, blood vessels or tissue to make them more visible. Depending on the type of contrast agent that is used, it may cause decreased kidney function or worsen kidney function in people who already have decreased kidney function. Therefore, we will monitor your kidney function closely while you participate in this study. If there is any change in your kidney function, we may have to remove you from the study.

Uncommonly, some people have allergic reactions (such as hives and itching) to the contrast agent. Serious reactions (for example, drop in blood pressure, difficulty breathing or severe allergic reaction and death) are rare.

#### Reproductive Risks:

The drug used in this research study may affect a fetus. While participating in this research study and for 4 months after, you should not become pregnant or father a baby, and should not nurse a baby. We can provide counseling about preventing pregnancy for either male or female study participants. Let your doctor know immediately if you become pregnant or find out that you are going to be the father of a child.

#### Non-Physical Risks:

Because of side effects or the time required for tests and clinic visits while you are on this research study, you may be unable to keep up with your normal daily activities.

## G. WHAT ARE THE BENEFITS OF THE RESEARCH STUDY?

We do not know if taking part in this study will help you. This study may help researchers learn information that could help people in the future.

## H. CAN I STOP BEING IN THE RESEARCH STUDY AND WHAT ARE MY RIGHTS?

You have the right to choose not to sign this form. If you decide not to sign this form, you cannot participate in this research study.


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | - 55 Aug 19 |

| NCT number: NCT03279692 |
|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

You can stop being in the research study at any time. Tell the research doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop. Leaving the research study will not affect your medical care outside of the research study.

If you choose not to participate, are not eligible to participate, or withdraw from this research study, this will not affect your present or future care and will not cause any penalty or loss of benefits to which you are otherwise entitled.

It is important to tell the research doctor if you are thinking about stopping so your research doctor can evaluate the risks from stopping the drug. Another reason to tell your research doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

#### I. WILL I BE PAID TO TAKE PART IN THIS RESEARCH STUDY?

You will not be paid for participating in this study.

We may use your samples and information to develop a new product or medical test to be sold. The sponsor and hospital may benefit if this happens. There are no plans to pay you if your samples are used for this purpose.

## J. WHAT ARE THE COSTS?

Taking part in this research study might lead to added costs to you or your insurance company.

You will not be charged for pembrolizumab. It is possible that pembrolizumab may not continue to be supplied free for some reason. If this would occur, your research doctor will talk with you about your options.

You or your insurance company will be charged for portions of your care during this research study that are considered standard care. You may be responsible for co-payments and deductibles that are typical for your insurance coverage.

If you have questions about your insurance coverage, or the items you might be required to pay for, please call financial services for information. The contact information for financial services are:

#### 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | VVC) 5-88 (Mc), WI |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

- Brigham and Women's Hospital: (617) 732-5524 or (617) 732-7485
- Dana-Farber Cancer Institute: (617) 632-3455
- Massachusetts General Hospital: (617) 726-2191

The National Cancer Institute provides an online resource to help people participating in cancer clinical trials understand which services their insurance company is required by law to pay. This can be found at the website below or can be provided by the study team:

www.cancer.gov or 1-800-4-CANCER (1-800-422-6237)

# K. WHAT HAPPENS IF I AM INJURED OR BECOME SICK BECAUSE I TOOK PART IN THIS RESEARCH STUDY?

If you think you have been injured as a result of taking part in this research study, tell the person in charge of this research study as soon as possible. The research doctor's name and phone number are listed in this consent form.

The treating hospital will offer you the care needed to treat injuries directly resulting from taking part in this research. These treatments will be billed to your insurance company. You will be responsible for deductibles and co-payments. There are no plans to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

We will need to collect certain personal information about you for insurance or payment reporting purposes, such as your name, date of birth, gender, social security number or Medicare identification number and information related to this research study. We may be required to report this information to the Centers for Medicare & Medicaid Services. We will not use this information for any other purpose.

# L. WHAT ABOUT CONFIDENTIALITY?

We will take measures to protect the privacy and security of all your personal information, but we cannot guarantee complete confidentiality of study data.

Medical information created by this research study may become part of your hospital medical record and may be forwarded to your primary doctor.


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | 5000 500000 5000 5000000 |

3/28/2023 4:35 PM

| NCT number: NCT03279692 | |
|-------------------------|---|
| | _ |

#### Research Consent Form for Biomedical Research

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

Information that does not become part of your medical record will be stored in your study file. It may also become part of a DF/HCC research database.

The results of this research study may be published. You will not be identified in publications without your permission.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## M. WHOM DO I CONTACT IF I HAVE QUESTIONS ABOUT THE RESEARCH STUDY?

If you have questions about the study, please contact the research doctor or study staff as listed below:

#### **Massachusetts General Hospital**

Priscilla Brastianos, MD: (617) 724-8770

## **Dana-Farber Cancer Institute**

• Eudocia Karem Quant Lee, MD, MPH: (617) 632-2166

**24-hour contact**: Please contact Massachusetts General Hospital at 617-724-4000 and ask that your doctor be paged.

For questions about your rights as a research participant, please contact a representative of the Office for Human Research Studies at Dana-Farber Cancer Institute (617) 632-3029. This can include questions about your participation in the study, concerns about the study, a research related injury, or if you feel/felt under pressure to enroll in this research study or to continue to participate in this research study.

# N. FUTURE USE OF DATA AND SPECIMENS

Your personal information and/or biospecimens collected during this study may be stored and used for future research. If so, any personal identifiers will be removed so that the information or samples cannot be linked back to you. As a result, we will no longer be able to identify and destroy them.


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | A-85 |

| 8/28/2023 4:35 PM | NC. |
|-------------------|-----|

NCT number: NCT03279692

#### Research Consent Form for Biomedical Research

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

Investigators, including investigators from collaborating institutions, can request this data and samples for new research. Samples and data may also be shared with outside non-profit academic investigators as well as with for-profit pharmaceutical investigators or commercial entities, with whom we collaborate

You will not be asked to provide additional informed consent for the use of your de-identified information or samples in future research.

Future research studies may include genetic research. Your genes are unique to you. At this time, you cannot be identified through this research. There is a risk that you might be reidentified in the future as genetic research progresses.

#### O. PRIVACY OF PROTECTED HEALTH INFORMATION

Federal law requires Dana-Farber/Harvard Cancer Center (DF/HCC) and its affiliated research doctors, health care providers, and physician network to protect the privacy of information that identifies you and relates to your past, present, and future physical and mental health conditions ("protected health information"). If you enroll in this research study, your "protected health information" will be used and shared with others as explained below.

## 1. What protected health information about me will be used or shared with others during this research?

- Existing medical records, including mental health records.
- New health information created from study-related tests, procedures, visits, and/or questionnaires

# 2. Why will protected information about me be used or shared with others?

The main reasons include the following:

- To conduct and oversee the research described earlier in this form:
- To ensure the research meets legal, institutional, and accreditation requirements;
- To conduct public health activities (including reporting of adverse events or situations where you or others may be at risk of harm); and


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | 5000 5000 5000 5000 |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

- To provide the study sponsor with information arising from an adverse event or other event that relates to the safety or toxicity of the drug(s) used in the study and for the purpose of this or other research relating the study drug(s) and their use in cancer;
- To better understand the diseases being studied and to improve the design of future studies; and,
- Other reasons may include for treatment, payment, or health care operations. For example, some medical information produced by this research study may become part of your hospital medical record because the information may be necessary for your medical care. (You will also be given a notice for use and sharing of protected health information.)

#### 3. Who will use or share protected health information about me?

 DF/HCC and its affiliated research doctors and entities participating in the research will use and share your protected health information. In addition, other DF/HCC offices that deal with research oversight, billing or quality assurance will be able to use and share your protected health information.

# 4. With whom outside of DF/HCC may my protected health information be shared?

While all reasonable efforts will be made to protect the confidentiality of your protected health information, it may also be shared with the following entities:

- Outside individuals or entities that have a need to access this information to perform functions relating to the conduct of this research such as analysis by outside laboratories on behalf of DF/HCC and its affiliates (for example, data storage companies, insurers, or legal advisors).
- The sponsor of the study, its subcontractors, representatives, business partners, and its agent(s): DF/HCC
- The funder of the study, its subcontractors, representatives, business partners, and its agent(s): Merck
- Other research doctors and medical centers participating in this research, if applicable
- Federal and state agencies (for example, the Department of Health and Human Services, the Food and Drug Administration, the National Institutes of Health, and/or the Office for Human Research Protections), or other domestic or foreign government bodies if required by law and/or

| Page 14 | of 18 |
|---------|-------|
|---------|-------|

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center
BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

necessary for oversight purposes. A qualified representative of the FDA and the National Cancer Institute may review your medical records.

- Hospital accrediting agencies
- A data safety monitoring board organized to oversee this research, if applicable

Some who may receive your protected health information may not have to satisfy the privacy rules and requirements. They, in fact, may share your information with others without your permission.

#### 5. For how long will protected health information about me be used or shared with others?

 There is no scheduled date at which your protected health information that is being used or shared for this research will be destroyed, because research is an ongoing process.

### 6. Statement of privacy rights:

- You have the right to withdraw your permission for the research doctors and participating DF/HCC entities to use or share your protected health information. We will not be able to withdraw all the information that already has been used or shared with others to carry out related activities such as oversight, or that is needed to ensure quality of the study. To withdraw your permission, you must do so in writing by contacting the researcher listed above in the section: "Whom do I contact if I have questions about the research study?"
- You have the right to request access to your protected health information that is used or shared during this research and that is related to your treatment or payment for your treatment, but you may access this information only after the study is completed. To request this information, please contact the researcher listed above in the section: "Whom do I contact if I have guestions about the research study?"

#### 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | 5000 500000 5000 5000000 |

| 8/28/2023 4:35 PM | NCT number: NCT03279692 |
|-------------------|-------------------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

#### P. DOCUMENTATION OF CONSENT

My signature below indicates:

- I have had enough time to read the consent and think about participating in this study;
- I have had all of my questions answered to my satisfaction;
- · I am willing to participate in this study;
- I have been told that my participation is voluntary and I can withdraw at any time

| Signature of Participant or Legally Authorized Representative | Date |
|---|---|
| Relationship of Legally Authorized Repre | esentative to Participant |


| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | 5000 5000 5000 5000 |

| NCT number: NCT03279692 |
|-------------------------|

Dana-Farber/ Harvard Cancer Center BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates

OHRS 02.03.2017

# To be completed by person obtaining consent: **Adult Participant**

| The consent discussion was initiated on (date). |
|---|
| Signature of individual obtaining consent: |
| Printed name of above: |
| Date: |
| <ul> <li>A copy of this signed consent form will be given to the participant or legally authorized<br/>representative.</li> </ul> |
| 1) The participant is an adult and provided consent to participate. |
| 1a) Participant (or legally authorized representative) is a non-English speaker and<br>signed the translated Short Form in lieu of English consent document: |
| As someone who understands both English and the language spoken by the participant, I interpreted and/or witnessed, in the participant's language, the researcher's presentation of the English consent form. The participant was given the opportunity to ask questions. |
| Signature of Interpreter/Witness: |
| Printed Name of Interpreter/Witness: |
| Date: 1b) Participant is physically unable to sign the consent form because: |
| ☐ The participant is illiterate. |
| ☐ The participant has a physical disability. |
| Other (please describe): |
| The consent form was presented to the participant who was given the opportunity to ask questions and who communicated agreement to participate in the research. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |
| 2) The participant is an adult who lacks capacity to provide consent and his/her legally<br>authorized representative: |
| Page 17 of 19 |

#### 

| DFCI Protocol Number: 17-296 | Approved Date (DFCI IRB Approval): 01/24/2023 |
|---|---|
| Date Posted for Use: 03/14/2023 | - 50 Oct. 100 Oct. 10 |

| 3/28/2023 4:35 PM | NCT number: NCT03279692 | |
|---|---|---|
| Research Consent Form | | |
| for Biomedical Research | | |
| Dana-Farber/ Harvard Cancer C | enter | |
| BIDMC/BCH/BWH/DFCI/MGH/Partners Network Affiliates | | OHRS 02.03.2017 |
| 2a) gave permission | for the adult participant to participate | |

☐ 2b) did not give permission for the adult participant to participate